CLINICAL TRIAL: NCT02996201
Title: Electronic Patient Reporting of Side Effects to Chemotherapy Among Breast Cancer Patients Using the Patient-Reported Outcomes Version of Common Terminology Criteria for Adverse Events (PRO-CTCAE): A Cluster Randomized Controlled Trial
Brief Title: Electronic Patient Reporting of Side Effects to Chemotherapy: A Cluster Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Helle Pappot, Chief physician, Rigshospitalet, Denmark
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R113-A7084-14-S34
Record Dates: First submitted 2016-11-04; First posted 2016-12-19 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Adverse Event; Cancer, Breast; Chemotherapeutic Toxicity; Patient Outcomes Assessments
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic reporting of PRO-CTCAE items (Experimental): Patients report PRO-CTCAE symptoms on a tablet computer before each cycle of chemotherapy
  Interventions: Other: Completion of PRO-CTCAE items before consultation
- Standard practice (No Intervention)

INTERVENTIONS:
Other: Completion of PRO-CTCAE items before consultation — Patients report PRO-CTCAE symptoms on a tablet computer before each cycle of chemotherapy
  Arms: Electronic reporting of PRO-CTCAE items

SUMMARY:
The aim of this study is to determine whether the use of breast cancer patients' own electronic reporting of side effects to chemotherapy in a treatment setting has an impact on the handling of side effects and on the number of hospitalizations, febrile neutropenia and dose adjustments. We are using the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) for the patients' reporting of side effects.

ELIGIBILITY:
Gender •Female: only female participants are being studied

Minimum age

•18 years

Maximum age •N/A

Accepts Healthy Volunteers

•No

Eligibility Criteria

Inclusion criteria

* Breast cancer patients starting adjuvant chemotherapy in the period November 1, 2015 - September 1, 2016 in Danish oncology clinics

Exclusion Criteria:

* More than six scheduled cycles of chemotherapy
* Not able to read and understand Danish language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Dose adjustments reported in the medication treatment sheet before each cycle of chemotherapy (5 time points with three weeks interval) | up to 18 weeks of treatment in the period betweeen November 1, 2015 and January 31, 2017

SECONDARY OUTCOMES:
Number of hospitalizations reported in the medical record after each of the six cycles of chemotherapy | up to 18 weeks of treatment in the period betweeen November 1, 2015 and January 31, 2017
Febrile neutropenia reported in the medical record after each of the six cycles of chemotherapy | up to 18 weeks of treatment in the period betweeen November 1, 2015 and January 31, 2017
Detailed description of side effects in the medical record before start of chemotherapy and after each six cycles of chemotherapy | up to 18 weeks of treatment in the period betweeen November 1, 2015 and January 31, 2017
Handling of side effects documented in the medical record | up to 18 weeks of treatment in the period betweeen November 1, 2015 and January 31, 2017
Patients' experience of communication and handling of side effects measured in questionnaire survey and qualitative interviews | up to18 weeks of chemotherapy in the period November 1, 2015 - January 31, 2017
Patient and staff compliance as registerede by the software used | up to 18 weeks (November 1, 2015 - January 31, 2017)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pappot H, Baeksted CW, Nissen A, Knoop A, Mitchell SA, Christensen J, Hjollund NH, Johansen C. Clinical effects of assessing electronic patient-reported outcomes monitoring symptomatic toxicities during breast cancer therapy: a nationwide and population-based study. Breast Cancer. 2021 Sep;28(5):1096-1099. doi: 10.1007/s12282-021-01244-x. Epub 2021 Apr 9. PMID 33837509
- [Derived] Baeksted CW, Nissen A, Knoop AS, Pappot H. Patients' experience of communication and handling of symptomatic adverse events in breast cancer patients receiving adjuvant chemotherapy. Res Involv Engagem. 2019 Nov 20;5:36. doi: 10.1186/s40900-019-0171-1. eCollection 2019. PMID 31832240